CLINICAL TRIAL: NCT06714656
Title: Drivers and Barriers for Adopting Healthy and Sustainable Food Swaps in Young. The FOOD SWAPS Study
Brief Title: Drivers and Barriers for Adopting Healthy and Sustainable Food Swaps in Young
Acronym: FOOD-SWAPS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aberdeen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: FOOD-SWAPS
Record Dates: First submitted 2024-11-22; First posted 2024-12-03 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Diet Modification; Sustainable Food Consumption
Keywords: diet; sustainable food choices; food swaps; N of 1 study

STUDY DESIGN:
Intervention Model Description: The study will be conducted as a 24-week (~ 6 months) interventional N-of-1 study with an A1-B-A2 design (8 weeks per study arm). The first A-period represents an observational phase, the B-period represents an intervention phase with personalised food swaps and dietary advice on how to incorporate these swaps into the diet, and the second A-period represents an observational/follow-up period.
Masking Description: This will have an N of 1 design and will not be randomised.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- N of 1 intervention (Experimental): Personalised food swaps and dietary advice on how to incorporate these swaps into the diet
  Interventions: Other: Food Swap

INTERVENTIONS:
Other: Food Swap — Personalised food swaps and dietary advice on how to incorporate these swaps into their usual diet

SUMMARY:
Food represents one of the greatest health and environmental challenges of the 21st century. Consuming less of the most environmentally damaging foods, such as meat, is considered an effective method to reduce food-related greenhouse gas emissions. The aim of these N-of-1 FOOD SWAP intervention studies is to investigate whether and which physiological, psychological and environmental factors, at an individual level, modify the adoption and adherence of food swaps aiming to reduce the intake of red meat and replace this with fish or plant-based foods, in young adults. The series of N-of-1 studies will also assess whether an 8-week food swap intervention will improve general health markers such as blood pressure, plasma lipids and glucose, and blood/urinary metabotype. This approach will provide insight into physiological, behavioural and environmental factors that can help explain individual fluctuations in adherence and physiological outcomes common in nutrition studies. In the future, this should enable us to tailor how we deliver effective individualised interventions and better consider and control for factors affecting adherence and response to dietary interventions.

DETAILED DESCRIPTION:
In the past 50 years, there has been a shift towards unhealthy diets high in calories and heavily processed and animal-based foods. Transitions to unhealthy diets are increasing the burden of obesity and diet-related non-communicable diseases and contribute to environmental degradation. Dietary guidelines are an important behaviour change policy tool to guide consumers regarding foods and diets. However, healthy diets alone may not produce substantial reductions in greenhouse gas emissions; therefore, dietary guidelines need to include recommendations for environmental sustainability. Thus far, only a few countries have started to produce dietary recommendations for health based on nutrient requirements, but which also aim to reduce environmental impact by decreasing the intake of specific foods like meat and dairy. However, dietary guidelines in most countries fail to consider the reasons behind people food choices, such as habits, preferences, affordability, circumstance, culture and social norms.

Food purchasing is a key behavioural precursor to food consumption, and interventions targeting the nutritional and environmental quality of food prior to or during shopping present a clear opportunity for effective behaviour change. Interventions implemented in grocery stores, particularly those that manipulate price, suggest that food swaps, and perhaps manipulating item availability, impact purchasing and could play a role in public health strategies to improve health. Using swaps to promote health would be a scalable and low-cost intervention, but currently, there is limited evidence of its effectiveness. The success of offering swaps depends on consumers adopting the suggested swaps, but most studies thus far have not explored why swap acceptance rates could be low. Acceptance could be low due to how swaps were framed, perceived to restrict freedom and personal autonomy, and perceived to be less palatable. Also, many consumers put lower importance on health messages and higher importance on taste and price. Indeed, product costs have been a particularly crucial factor for those on lower incomes, and lower prices can encourage choices of healthier products more effectively than health status labels.

A change towards healthier, more environmentally sustainable and affordable diets is feasible in population-level studies across European populations. Yet dietary intakes are hugely variable across income groups, age groups, and groups defined by other demographics; therefore, individual/group behavioural change may vary from the general population-level solutions.

From a consumer perspective, reducing food waste, consuming fewer calories, and consuming less environmentally damaging foods (meat and dairy) are the most effective methods to reduce food-related greenhouse gas emissions. The EAT-Lancet Commission concluded that there needs to be a greater than 50% reduction in global red meat consumption, among other dietary changes, to achieve a sustainable, healthy food system, whilst, in the UK, it has been suggested that beef consumption needs to decrease by 89% to stay within planetary boundaries. In 2010, the Scientific Advisory Committee on Nutrition (SACN) recommended that UK adults with high intakes of red and processed meat (>90 grams per day) should reduce their intake to a maximum of 70 grams per day (the average red and processed meat consumption of adult consumers at that time: 88 grams per day for men and 52 grams per day for women), which was mainly based on the relationship between red meat and processed meat intake and colorectal cancer. More recently, in 2020, the UK Committee on Climate Change (CCC) advised that consumption of all meat and dairy should fall by at least 20% by 2030, and that consumption of all meat should fall by at least 35% by 2050, to reduce our food system-based carbon footprint significantly. In 2023, the Scottish Government partially accepted this recommendation.

Globally, average per capita meat consumption is increasing, driven by population growth, rising incomes, and socio-cultural traditions that place a high value on eating meat. However, whilst per capita meat consumption is high in the UK, it is beginning to decline: from 2008 to 2019, average total meat consumption per capita per day decreased from 104 to 86 grams, including an absolute reduction in red meat consumption of 14 grams, an absolute reduction in processed meat consumption of 7 grams, and an increase in white meat consumption of 3 grams. Attitudes towards meat consumption and meat reduction differ between subgroups of the population, and therefore, individual-level interventions, such as tailored dietary advice, information, self-monitoring and personalised feedback, may represent a more effective behaviour change technique than general dietary guidelines.

In this study, red meat consumption behaviours will be monitored before, during and after an intervention that provides personalised food swaps to:

i) reduce individual intake of red meat (including beef, veal, lamb, and pork), by 20% (following the recommendation of the Climate Change Committee, but targeting the consumption of red meat rather than total meat), or ii) reduce the individual intake of red meat to 60 grams per day, or 420 grams per week, or 240 grams per 4 days (following SACN advice, but taking into account that the average per capita intake of red and processed meat has come down from 70 grams per day 10 years ago) in a target population of young adults with a high intake of red meat, either fresh or processed ( less than 70 grams per day or 280 grams per 4 days), depending on each participant's preference.

Food swaps will include fish or plant-based foods, not white meat. To establish individual drivers and barriers to adopting such food swaps, there is a need to be able to see what behavioural, physiological and environmental factors unique to each participant co-occur with or predict changes in the uptake of recommended food swaps. This will provide a greater understanding of what personal factors affect adherence. Through an N-of-1 design, behavioural and environmental factors can be measured in real-time via Ecological Momentary Assessment (EMA), minimising retrospective recall bias. EMA is easily combined with technology such as smartphones and wrist devices such as the m-Path or PRO-Diary device (see below) to deliver time-stamped questionnaires to participants.

ELIGIBILITY:
Inclusion Criteria:

* men and women
* aged 18-30 years,
* having a high baseline consumption of red meat (More than 70 grams per day or 280 grams per 4 days)
* who are willing to make their diet healthier and more sustainable but do not know how or are facing barriers

Exclusion Criteria:

* Having a lower red meat consumption (less than 70 grams per day or 240 grams per 4 days)
* being vegetarian or vegan
* having a clinical diagnosis of hypertension or high cholesterol, having unstable or untreated thyroid disorder
* taking blood pressure and/or cholesterol-lowering medications (e.g. beta blockers or statins)
* having food allergies, being on a weight loss diet or having lost >5kg in the last 6 months
* having a history of an eating disorder.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-12-09 (Actual); Primary Completion 2027-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Grams of red meat consumption | 6 months
  During the first eight weeks (period A1), participants will be instructed to follow their usual diet. From week 9 (period B), participants will start the intervention, where they will receive the food swaps identified and agreed by them during a food swap interview. During the final eight weeks (period A2), participants will cease intervention products. The grams of red meat will be monitored before, during and after the intervention.

SECONDARY OUTCOMES:
Weight | 6 months
  Kg of bodyweight
Nutiritional status | 6 months
  Body Mass Index
Blood pressure | 6 months
  Including systolic pressure and diastolic pressure readings (mmHg)
Total cholesterol | 6 months
  mmol/L, measured every 4 weeks
Fasting blood glucose | 6 months
  mg/dL, measured every 4 weeks
urinary metabotype | 6 months
  Masured at the start and the end of the intervention period B.

CONTACTS AND LOCATIONS:
Overall Officials: Baukje de Roos, Professor, Principal Investigator — UoA
Locations (1):
- The Rowett Institute, University of Aberdeen, Aberdeen, United Kingdom

IPD SHARING:
Plan to Share IPD: No